CLINICAL TRIAL: NCT02981810
Title: Evaluation of Coblation Channeling Treatment for Chronic Tonsillitis.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Principal Investigator, Itzhak Braverman, Assitant Proffessor, Hillel Yaffe Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0046-16-HYMC
Record Dates: First submitted 2016-11-13; First posted 2016-12-05 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2016-12

CONDITIONS: Chronic Tonsillitis
Keywords: TONSILLAR COBLATION
MeSH Terms: interventions — Tonsillectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- control (Active Comparator): tonsillectomy
  Interventions: Procedure: tonsillectomy
- coblation (Experimental): coblation of the tonsills
  Interventions: Device: Arthrocare® Corporation (ArthroCare Corporation, 7500 Rialto Boulevard Austin, Texas 78735) COBLATION electrode ReFlex Ultra 55*

INTERVENTIONS:
Device: Arthrocare® Corporation (ArthroCare Corporation, 7500 Rialto Boulevard Austin, Texas 78735) COBLATION electrode ReFlex Ultra 55* — The treatment was conducted using an Arthrocare® Corporation (ArthroCare Corporation, 7500 Rialto Boulevard Austin, Texas 78735) COBLATION electrode ReFlex Ultra 55* for tonsillar tissue ablation at low temperatures with only one treatment. All the patients underwent tonsil channeling treatment with coblation, and 4-6 channels were done in each tonsil under local anesthesia, in the operating room. The patients were observed overnight.
  Arms: coblation
Procedure: tonsillectomy
  Arms: control

SUMMARY:
To evaluate coblation channeling treatment for chronic tonsillitis. Does Tonsillar ablation can create changing in the tonsillar medium for recurrent tonsillar infections and stop the recurrent infections?

DETAILED DESCRIPTION:
The palatine tonsil consists of an epithelial crypt (invaginated pocket) surrounded by dense clusters of lymph nodules, each with a germinal center where lymphocytes proliferate. The nodules are embedded in a mass of diffuse lymphoid tissue that consists of lymphocytes migrating to and from the germinal centers.

Increasing the surface area of the crypts is one way to facilitate the contact of antigens (bacteria) with the immune cells. The epithelium may specialize to form an openmeshwork of cells which allows the infiltration of the epithelium by lymphocytes and macrophages. Tonsillar lymphoid nodules consist mainly of B-lymphocytes. Other areas are occupied by T-lymphocytes, activated B-lymphocytes and other cells of the immune system. Inside the crypts, where cells of the immune system often invade the epithelium, it will be difficult to find the specific boundary between epithelium and lymphoid tissue. The bacterial material and biofilms1 sits in crypts and may start a new infection from time to time. The epithelium lining the crypt corresponds with that on the adjacent surface - stratified squamous in the tongue and palate or pseudo stratified columnar in the pharynx. In either case, the epithelium may be heavily infiltrated with lymphocytes, and the crypt may be filled with lymphocytes and other debris.

The tonsillar crypts have an important role in chronic tonsillitis. They are covered by stratified epithelium and may be initiated via the epithelium to mount immune responses to various presenting antigens. Go M. et al, investigated the expression and function of tight junctions in the epithelium of human palatine tonsils from patients with tonsillar hypertrophy or recurrent tonsillitis. These studies suggested unique expression of tight junctions in human palatine tonsillar epithelium, and it was suggested that the crypt epithelium may possess an epithelial barrier different from that of the surface epithelium2.

Bacteria within biofilms are resistant to host defenses and antibiotics. The presence of bacterial biofilms within the tissue and crypts of inflamed tonsils may explain the chronic and recurrent characteristics of some forms of tonsillitis. There is strong anatomical evidence for the presence of bacterial biofilms in chronically diseased tonsils1. Using a novel visualization approach in single sections of human mucosal tissue, the presence of biofilms was demonstrated on tonsils in most (17/24 [70.8%]) patients with tonsillitis3.

One study investigated the difference in follicle size and numbers in tonsils for patients with tonsillar hypertrophy and recurrent tonsillitis using an image analysis method. There was no significant difference in the mean follicle numbers per counting field between recurrent tonsillitis and tonsillar hypertrophy. However, they demonstrated that tonsillar hypertrophy is characterized histologically by an enlargement of follicles compared with recurrent tonsillitis, indicating a hyperplastic condition of lymphoid cells in the germinal centers. It may also explain the difference in etiology and immune mechanism between tonsillar hypertrophy and recurrent tonsillitis4.

Coblation is a non-heat driven process in which radiofrequency energy is applied to a conductive medium (usually saline) causing a highly focused plasma field to form around the electrodes. The plasma field is comprised of highly ionized particles. These ionized particles have sufficient energy to break organic molecular bonds within tissue. Instead of exploding tissue, coblation causes a low-temperature molecular disintegration, resulting in minimal tissue damage to surrounding areas.

A novel treatment for chronic tonsillitis is now suggested by the inventors, this method being based on treating the source of recurrent bacterial infections in the tonsillar tissue, specifically the tonsillar crypts.

By treatment of the crypts and tonsillar tissue it may be possible to decrease the possible antigen-immune system interaction and inflammation.

Without being bound to a specific theory, it is suggested that the combination of the radio frequency energy and the fluid creates a "plasma" field containing highly ionized particles, which have sufficient energy to break organic molecular bonds that can remove tissue selectively without excessive heat production and damage the surrounding tissue.

Material and Methods

The study protocol was approved by the The Hillel Yaffe Medical Center's Ethics and Helsinki Committee.

60 patients suffering from chronic tonsillitis will be treated by Coblation channeling to the tonsils.

The treatment was conducted using an Arthrocare® Corporation (ArthroCare Corporation, 7500 Rialto Boulevard Austin, Texas 78735) COBLATION electrode ReFlex Ultra 55* for tonsillar tissue ablation at low temperatures with only one treatment. All the patients underwent tonsil channeling treatment with coblation, and 4-6 channels were done in each tonsil under local anesthesia, in the operating room. The patients were observed overnight.

A control group included 60 patients with chronic tonsillitis with indication for tonsillectomy will underwent tonsillectomy.

The patients selected are older than 18 years old, and were healthy, without any chronic diseases other than chronic tonsillitis. Diagnosis of chronic tonsillitis was based on history and medical examination. The criteria were: 1. At least 4 occasions of tonsillitis in the last year that were treated (positive throat swab for Streptococci Group A will contribute towards the diagnosis). 2. Recurrent or chronic throat pain. 3. Hypertrophic tonsils of chronic tonsillitis. Patients that were not included: 1. Disease of the mouth or pharyngeal mucosa-like ulcers. 2. Allergy to drugs. 3. Gastrointestinal reflux. 4. Any contraindication for tonsillectomy. 5. Peritonsillar abscess in the past.

Final evaluations were by follow-up of the patients 1,2,4,6 and 12 months after the beginning of treatment. At each visit, evaluation of the treatment was done by investigating the degree of throat pain or tonsillitis after the treatment, number of tonsillitis per year, examination of the tonsils, post treatment pain score by VISUAL-ANALOG-SCALE (VAS) SCORES. The following parameters were recorded: the size of tonsils before and after treatment, number of occurrences of tonsillitis after one year, and if there was any post-treatment bleeding.

The results will be statistically evaluated .

ELIGIBILITY:
Inclusion Criteria:

* Patients without any chronic diseases other than chronic tonsillitis. Diagnosis of chronic tonsillitis is based on history and medical examination. The criteria are: 1. At least 3 occasions of tonsillitis in the last year that were treated (positive throat swab for Streptococci Group A will contribute towards the diagnosis). 2. Recurrent or chronic throat pain. 3. Hypertrophic tonsils of chronic tonsillitis.

Exclusion Criteria:

* Disease of the mouth or pharyngeal mucosa-like ulcers.
* Allergy to drugs.
* Gastrointestinal reflux.
* Peritonsillar abscess in the past.
* Pregnant women
* Oncologic patients
* Hematologic disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-12; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Change in the number of visits at the doctor due to throat pain- using a questionnaire | 12 months
  the patient will be asked to report in specific time points in his/hers follow up: after 1 month, 2months, 4 months, 6 months and 12 months
Change in the number of antibiotic treatment was indicated after the procedure- using a questionnaire | 12 month
  the patient will be asked to report in specific time points in his/hers follow up: after 1 month, 2months, 4 months, 6 months and 12 months
questionnaires to subjectively evaluate the change in patient's discomfort while swallowing | 12 month
  the patient will be asked to report in specific time points in his/hers follow up: after 1 month, 2months, 4 months, 6 months and 12 months
visual documentation of the pharynx with video camera | 12 month

SECONDARY OUTCOMES:
post operative pain assessment via VAS (VISUAL ANALOG SCALE) scores | up to 7 days
location and amount of bleeding- post surgical documentation | up to 7 days

IPD SHARING:
Plan to Share IPD: Undecided